CLINICAL TRIAL: NCT01657487
Title: Comparing Treatment Efficacy With High and Medium Dose of Fluticasone in Combination With Salmeterol in COPD Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Collaborators: Research Ethics Review Committee (Ambiguous)
Responsible Party: Principal Investigator, Shih-Lung Cheng, Division of Pulmonary Medicine, Department of Internal Medicine, Far Eastern Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 099013-F
Record Dates: First submitted 2012-08-02; First posted 2012-08-06 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Percentage of Annual Acute Exacerbation; Quality of Life
Keywords: COPD; Fluticasone/Salmeterol; high dose
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone; Salmeterol Xinafoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fluticasone/salmeterol high dose (Experimental): COPD patients treating with high dose of ICS (Fluticasone 1000ug/day) combined with Salmeterol (25ug/day)
  Interventions: Drug: Fluticasone/Salmeterol high dose
- Fluticasone/Salmeterol medium dose (Active Comparator): COPD patients treating with medium dose of ICS (Fluticasone 500ug/day) combined with Salmeterol (25ug/day)
  Interventions: Drug: Fluticasone/Salmeterol high dose

INTERVENTIONS:
Drug: Fluticasone/Salmeterol high dose
  Other Names: COPD patients treating with high dose of ICS (Fluticasone 1000ug/day) combined with Salmeterol (25ug/day)

SUMMARY:
This study is to investigate and compare treatment efficacy with high and medium dose of fluticasone in combination with salmeterol in COPD patients.

DETAILED DESCRIPTION:
Diagnosis and criteria for inclusion and exclusion:

Inclusion:

1. Male or female outpatients aged 40 years≧
2. Current or ex-smoker, with smoking history 10 pack≧- years
3. COPD (FEV1/FVC < 70%) patients with post-bronchodilator FEV1 70% ≦predicted value, without bronchial reversibility (10% increase post ≦bronchodilator)

Exclusion:

1. Diagnosis or suspicion of sleep apnea.
2. Concurrent rhinitis, eczema, and asthma.
3. Clinically overt bronchiectasis, lung cancer, active tuberculosis, or other known specific pulmonary disease.
4. A chest X-ray indicating diagnosis other than COPD that might interfere with the study.
5. Major disease abnormalities are uncontrolled on therapy.
6. Alcohol or medication abuse.
7. Patients had lower respiratory tract infections or received systemic steroid in the 4 weeks prior to the commencement of study.
8. Unable or unwilling to comply with all protocol

Test product:

fluticasone125 mcg/salmetrol 25 mcg ( Seretide 125 Evohaler ) fluticasone250 mcg/salmetrol 25 mcg ( Seretide 250 Evohaler ) Formulation: fluticasone/salmeterol, 125/25 mcg/puff Dose: 2 puffs bid

ELIGIBILITY:
Inclusion Criteria:

1. Male or female outpatients aged 40 years≧
2. Current or ex-smoker, with smoking history 10 pack≧- years
3. COPD (FEV1/FVC < 70%) patients with post-bronchodilator FEV1 70% ≦predicted value, without bronchial reversibility (10% increase post ≦bronchodilator)

Exclusion Criteria:

1. Diagnosis or suspicion of sleep apnea.
2. Concurrent rhinitis, eczema, and asthma.
3. Clinically overt bronchiectasis, lung cancer, active tuberculosis, or other known specific pulmonary disease.
4. A chest X-ray indicating diagnosis other than COPD that might interfere with the study.
5. Major disease abnormalities are uncontrolled on therapy.
6. Alcohol or medication abuse.
7. Patients had lower respiratory tract infections or received systemic steroid in the 4 weeks prior to the commencement of study.
8. Unable or unwilling to comply with all protocol

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-09 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
The changes of lung function parameters, including post bronchodilation forced expiratory volume in first second (FEV1) and forced vital capacity (FVC), before and after treatment. | Lung function change in one year
  We will compare the lung function changed in COPD patients treating with different doses of Fluticasone (500 and 1000ug)

SECONDARY OUTCOMES:
Annual rate of acute exacerbations | percentage of acute exacerbation in one year
  1. Annual rate of acute exacerbations
  2. The number of use of rescue medication
  3. Annual incidence of community-acquired pneumonia
  4. The changes of Health-related quality of life assessed by questionnaire (CAT or SGRQ) before and after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, Taipei, Taiwan